CLINICAL TRIAL: NCT06176391
Title: Spinal Cord Stimulation for Vasospastic Angina Pectoris - a Prospective Study
Brief Title: SCS for Vasospastic Angina Vasospastic Angina Pectoris - a Prospective Study
Acronym: VAP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, Frank Wille, MD, Principal Investigator, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL79947.018.21
Record Dates: First submitted 2023-11-26; First posted 2023-12-19 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Angina Pectoris; Angiospastic
Keywords: ANOCA (Angina with Non-Obstructive Coronary Artery disease); Spinal Cord Stimulation; Angina Pectoris
MeSH Terms: conditions — Angina Pectoris | interventions — Spinal Cord Stimulation

STUDY DESIGN:
Intervention Model Description: Prospective pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- single (Other): Subjects are their own control
  Interventions: Device: Spinal Cord Stimulation

INTERVENTIONS:
Device: Spinal Cord Stimulation — Single lead placement in the posterior thoracic epidural space (T1-T4) connected to a subcutaneous battery
  Other Names: Dorsal Column Stimulation

SUMMARY:
According to the 2020 Dutch guideline on chest pain (AP) without obstructive coronary artery disease, 70% of female and 30% of male patients undergoing a coronary angiogram (CAG), have no obstructive coronary artery disease.In the majority of patients the complaints are based on vascular dysfunction, including epicardial vascular spasms. For patients who are refractory to drug treatment, spinal cord stimulation (SCS) can be a treatment option. SCS is used for the treatment of refractory neuropathic and ischaemic pain. In recent studies the use of SCS is proven for refractory angina pectoris, but the group with refractory vasospastic angina pectoris (rVSA) predominantly seen in women with invalidating impairment of quality of life, is overlooked, as no evidence of obstruction is found at CAG. With this pilot study the investigators hypothesize that SCS is effective in reducing the number and intensity of angina attacks, reducing nitrate use, reducing inhospital treatment and ER presentations, thereby reducing medical costs, and above all, increasing quality of life.

DETAILED DESCRIPTION:
Rationale:

Of the patients undergoing a coronary angiogram because of chest pain (AP), 67% of female and 33% of male patients have no obstructive coronary artery disease. In the majority of patients (59-89%) the complaints are based on vascular dysfunction, including epicardial vascular spasms (EVS). For patients who are refractory to drug treatment, spinal cord stimulation (SCS) can be a treatment option. SCS is used for the treatment of refractory neuropathic and ischaemic pain. In recent studies the use of SCS is proven effective for refractory angina pectoris, but the group with refractory vasospastic angina pectoris (rVSA), predominantly seen in women with invalidating impairment of quality of life, is overlooked, as no evidence of obstruction is found at CAG. With this study the investigators hypothesize that SCS is effective in reducing the number and intensity of angina attacks, reducing nitrate use, reducing inhospital treatment and ER presentations, thereby reducing medical costs, and above all, increasing quality of life.

Objective: the main objective of this study is to evaluate the clinical effects of SCS on the number and intensity of VSA attacks. Secondary objective is to objectivate the effects of SCS on coronary spasms during the provocative acetylcholine test, and assess medical costs, patient satisfaction and quality of life.

Study design: prospective study in two phases. Phase 1: evaluation of clinical effectiveness. Phase 2: evaluation of SCS on vascular spasms during acetylcholine provocation test.

Study population: 10 patients with refractory AP due to epicardial vascular spasms.

Intervention: implantation with a SCS device with one or two lead(s) in the epidural space of T1 to T4, active electrodes depending on mapping of the painfull area, under local anesthesia and sedation. Acetylcholine provocation test during coronary angiogram at 6 months.

Main study parameters/endpoints: primary endpoint is the Seattle Angina Questionnaire (SAQ) at month 1 and 3. Secundary endpoints are presentation at ER, estimated medical costs, and patient satisfaction measured on a 11 point Numeric Rating Scale and quality of life with the EQ5D at month 3, compared to baseline. Endpoints of the acetylcholine test are changes in coronary flow and coronary diameter compared to baseline.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: SCS is proven to be safe for neuropathic and ischaemic pain and is widely used in clinical practice. With the positive results of an ongoing clinical trial for refractory coronary angina, the investigators estimate the efficacy of SCS to be around 80-90% in reducing VSA attacks with 50% after 3 months and therefore very effective in otherwise refractory drug treatment regiments. Furthermore, baseline study parameters will be extracted from the routine questionnaires and during visits to the outpatient clinic.

Only in patients who specifically consent to it, an additional acetylcholine test 6 months after SCS implantation during coronary angiography (CAG) is performed. This is an additional coronary angiogram procedure under local anesthesia which potentially provokes VSA. Done by experienced personal this is a safe test with a complication risk of 0-0.7% for severe cardiac complications, comparable to coronary angiogram with functional flow reserve measurement.

A potential benefit for the participants is that SCS results in reduction of VSA attacks, reduction of nitrate use, less presentation at an ER, an improved quality of life, and acceptation as standard treatment.

ELIGIBILITY:
Inclusion Criteria:

* VSA is objectivated with a provocative acetylcholine test
* mentally competent and able to fill in the questionnaires
* refractory VSA defined as disabling chest pain with a maximum tolerated dosage of calcium antagonists, long acting nitrates, angiotensin converting enzyme inhibitors for a minimum of three months
* absence of obstructive coronary artery disease evident in a main coronary artery (diameter stenosis<50%, Instant Flow Reserve (IFR) >0.89, or Fractional Flow reserve (FFR) >0.80)
* able to use the remote control of the SCS system

Exclusion Criteria:

* inability to visit the outpatient department for the follow-up visits
* unable to provide informed consent
* myocardial infarction in the previous three months
* procedures like percutaneous coronary intervention (PCI) or coronary artery bypass grafting (CABG), nor instability of the clinical signs and symptoms of refractory angina in the previous three months
* implanted pacemaker or implantable cardioverter-defibrillator (ICD) incompatible with SCS
* indication for ongoing anticoagulation therapy
* pregnant women and those who are breastfeeding

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-01-02 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Seattle Angina Questionnaire (SAQ) | baseline (before implant) - 1 month after implant - 3 months after implant
  For patients with coronary artery disease, the Seattle Angina Questionnaire (SAQ) has emerged as the most commonly used measure of disease-specific health status to quantify patients' symptoms of angina and the extent to which their angina affects their functioning and quality of life.
  Scores of 0 to 30 translate to daily angina, 31 to 60 to weekly angina, 61 to 99 to monthly angina, and 100 to no angina.

SECONDARY OUTCOMES:
Euroquol Quality of Life questionnaire (EQ5D-5L) | baseline (before implant) -1 month after implant - 3 months after implant
  The EQ-5D-5L is a self-assessed, health related, quality of life questionnaire. The scale measures quality of life on a 5-component scale including mobility, self-care, usual activities, pain/discomfort, and anxiety/depression.
  The maximum score of 1 indicates the best health state, by contrast with the scores of individual questions, where higher scores indicate more severe or frequent problems. In addition, there is a visual analogue scale (VAS) to indicate the general health status with 100 indicating the best health status.
Patient satisfaction - Numeric Rating Scale (NRS) 0-10 | 1 month and 3 months after implant
  11-point Likert-type scale
Complications and side effects | through study completion, an average of 6 months
  Related to SCS
Acetylcholine provocation test during coronary angiogram | 6 months after implant
  Test to objectivate coronary spasms (compared to baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Markus Hollmann, MD, PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)

IPD SHARING:
Plan to Share IPD: Yes
In progress
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 6 months after closure of database for 3 years
Access Criteria: On request

REFERENCES:
- [Background] Deer TR, Mekhail N, Provenzano D, Pope J, Krames E, Leong M, Levy RM, Abejon D, Buchser E, Burton A, Buvanendran A, Candido K, Caraway D, Cousins M, DeJongste M, Diwan S, Eldabe S, Gatzinsky K, Foreman RD, Hayek S, Kim P, Kinfe T, Kloth D, Kumar K, Rizvi S, Lad SP, Liem L, Linderoth B, Mackey S, McDowell G, McRoberts P, Poree L, Prager J, Raso L, Rauck R, Russo M, Simpson B, Slavin K, Staats P, Stanton-Hicks M, Verrills P, Wellington J, Williams K, North R; Neuromodulation Appropriateness Consensus Committee. The appropriate use of neurostimulation of the spinal cord and peripheral nervous system for the treatment of chronic pain and ischemic diseases: the Neuromodulation Appropriateness Consensus Committee. Neuromodulation. 2014 Aug;17(6):515-50; discussion 550. doi: 10.1111/ner.12208. PMID 25112889
- [Background] Murphy DF, Giles KE. Dorsal column stimulation for pain relief from intractable angina pectoris. Pain. 1987 Mar;28(3):365-368. doi: 10.1016/0304-3959(87)90070-4. PMID 3494978
- [Background] Mannheimer C, Eliasson T, Augustinsson LE, Blomstrand C, Emanuelsson H, Larsson S, Norrsell H, Hjalmarsson A. Electrical stimulation versus coronary artery bypass surgery in severe angina pectoris: the ESBY study. Circulation. 1998 Mar 31;97(12):1157-63. doi: 10.1161/01.cir.97.12.1157. PMID 9537342
- [Background] Mobilia G, Zuin G, Zanco P, Di Pede F, Pinato G, Neri G, Cargnel S, Raviele A, Ferlin G, Buchberger R. [Effects of spinal cord stimulation on regional myocardial blood flow in patients with refractory angina. A positron emission tomography study]. G Ital Cardiol. 1998 Oct;28(10):1113-9. Italian. PMID 9834863
- [Background] Dejongste MJ. Efficacy, safety and mechanisms of spinal cord stimulation used as an additional therapy for patients suffering from chronic refractory angina pectoris. Neuromodulation. 1999 Jul;2(3):188-92. doi: 10.1046/j.1525-1403.1999.00188.x. No abstract available. PMID 22151207
- [Background] Lopshire JC, Zhou X, Dusa C, Ueyama T, Rosenberger J, Courtney N, Ujhelyi M, Mullen T, Das M, Zipes DP. Spinal cord stimulation improves ventricular function and reduces ventricular arrhythmias in a canine postinfarction heart failure model. Circulation. 2009 Jul 28;120(4):286-94. doi: 10.1161/CIRCULATIONAHA.108.812412. Epub 2009 Jul 13. PMID 19597055
- [Background] Liu Y, Yue WS, Liao SY, Zhang Y, Au KW, Shuto C, Hata C, Park E, Chen P, Siu CW, Tse HF. Thoracic spinal cord stimulation improves cardiac contractile function and myocardial oxygen consumption in a porcine model of ischemic heart failure. J Cardiovasc Electrophysiol. 2012 May;23(5):534-40. doi: 10.1111/j.1540-8167.2011.02230.x. Epub 2011 Dec 8. PMID 22151312
- [Background] Taylor RS, De Vries J, Buchser E, Dejongste MJ. Spinal cord stimulation in the treatment of refractory angina: systematic review and meta-analysis of randomised controlled trials. BMC Cardiovasc Disord. 2009 Mar 25;9:13. doi: 10.1186/1471-2261-9-13. PMID 19320999
- [Background] Andrell P, Yu W, Gersbach P, Gillberg L, Pehrsson K, Hardy I, Stahle A, Andersen C, Mannheimer C. Long-term effects of spinal cord stimulation on angina symptoms and quality of life in patients with refractory angina pectoris--results from the European Angina Registry Link Study (EARL). Heart. 2010 Jul;96(14):1132-6. doi: 10.1136/hrt.2009.177188. Epub 2010 May 18. PMID 20483898
- [Background] McNab D, Khan SN, Sharples LD, Ryan JY, Freeman C, Caine N, Tait S, Hardy I, Schofield PM. An open label, single-centre, randomized trial of spinal cord stimulation vs. percutaneous myocardial laser revascularization in patients with refractory angina pectoris: the SPiRiT trial. Eur Heart J. 2006 May;27(9):1048-53. doi: 10.1093/eurheartj/ehi827. Epub 2006 Mar 22. PMID 16554313
- [Background] Vervaat FE, van der Gaag A, van Suijlekom H, Botman CJ, Teeuwen K, Wijnbergen I. Improvement in quality of life and angina pectoris: 1-year follow-up of patients with refractory angina pectoris and spinal cord stimulation. Neth Heart J. 2020 Sep;28(9):478-484. doi: 10.1007/s12471-020-01422-0. PMID 32430654
- [Background] Gibbons RJ, Abrams J, Chatterjee K, Daley J, Deedwania PC, Douglas JS, Ferguson TB Jr, Fihn SD, Fraker TD Jr, Gardin JM, O'Rourke RA, Pasternak RC, Williams SV, Gibbons RJ, Alpert JS, Antman EM, Hiratzka LF, Fuster V, Faxon DP, Gregoratos G, Jacobs AK, Smith SC Jr; American College of Cardiology; American Heart Association Task Force on Practice Guidelines. Committee on the Management of Patients With Chronic Stable Angina. ACC/AHA 2002 guideline update for the management of patients with chronic stable angina--summary article: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Committee on the Management of Patients With Chronic Stable Angina). Circulation. 2003 Jan 7;107(1):149-58. doi: 10.1161/01.cir.0000047041.66447.29. No abstract available. PMID 12515758
- [Background] Suwaidi JA, Hamasaki S, Higano ST, Nishimura RA, Holmes DR Jr, Lerman A. Long-term follow-up of patients with mild coronary artery disease and endothelial dysfunction. Circulation. 2000 Mar 7;101(9):948-54. doi: 10.1161/01.cir.101.9.948. PMID 10704159
- [Background] Deer T, Slavin KV, Amirdelfan K, North RB, Burton AW, Yearwood TL, Tavel E, Staats P, Falowski S, Pope J, Justiz R, Fabi AY, Taghva A, Paicius R, Houden T, Wilson D. Success Using Neuromodulation With BURST (SUNBURST) Study: Results From a Prospective, Randomized Controlled Trial Using a Novel Burst Waveform. Neuromodulation. 2018 Jan;21(1):56-66. doi: 10.1111/ner.12698. Epub 2017 Sep 29. PMID 28961366
- [Background] Chakravarthy K, Kent AR, Raza A, Xing F, Kinfe TM. Burst Spinal Cord Stimulation: Review of Preclinical Studies and Comments on Clinical Outcomes. Neuromodulation. 2018 Jul;21(5):431-439. doi: 10.1111/ner.12756. Epub 2018 Feb 12. PMID 29431275